## Comparison of the Relationship Between Age and Serum Paraoxonase /Arylesterase Activity of Patients With Acute Coronary Syndrome Presenting to the Emergency Department

## Decrease in Paraoxonase Enzyme Level and Myocardial İnfarction

Decision of the Ethics Committee of Bezmialem University dated 09.10.2019 and numbered 20/9

## **Study Protocol and Statistical Analysis**

Patients with myocardial infarction will be identified. heart attack to be proved by angio result. patients will be tested for HDL and troponin levels. Blood samples to be used in the study will be taken from patients admitted to our hospital emergency department and included in the study in 2020. Blood samples from the control group are also routine to the same hospital it will be taken from healthy people who come in for a checkup. For control and determination of paraoxonase enzyme activity in the patient group, 1 gel 5 ml biochemistry tube will be taken, biochemistry tubes at 4400 rpm for 10 min, to be centrifuged the serums will be placed in flat tubes without gel (unadulterated), kept at ( - ) 20 degrees until analysis is done and delivered to the laboratory as soon as possible. Patients will be divided into groups according to paraoxonase activity results. The "oneway Anova" test will be used for statistical analysis. Analyses "SPSS Version.21" to be evaluated in the package program and significance level to be made based on  $\alpha = 0.05$